CLINICAL TRIAL: NCT06444191
Title: A Phase 1, Single-Center, Open-Label Study to Evaluate the Pharmacokinetics and Tolerability of Rilzabrutinib (PRN1008) in Japanese and Caucasian Healthy Male and Female Subjects
Brief Title: Pharmacokinetics (PK) of Rilzabrutinib (PRN1008) in Healthy Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Principia Biopharma, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKM17089; U1111-1260-4452 (Registry Identifier: ICTRP); PRN1008-023 (Other: Sanofi Identifier); PKM17089 (Other: Sanofi Identifier)
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Rilzabrutinib (Experimental)
  Interventions: Drug: Rilzabrutinib
- Cohort 2: Rilzabrutinib (Experimental)
  Interventions: Drug: Rilzabrutinib

INTERVENTIONS:
Drug: Rilzabrutinib — Rilzabrutinib tablet(s) administered orally

SUMMARY:
This is a single-dose and multiple doses study to assess the Pharmacokinetics (PK) of rilzabrutinib as well as to evaluate the tolerability of rilzabrutinib in Japanese and Caucasian Healthy Male and Female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Japanese subjects must have both biological parents and all four grandparents of Japanese ancestry and born in a Japanese country of origin.
* Caucasian subjects must have four Caucasian grandparents (Hispanics of white race can be considered Caucasian).
* Healthy adult male or non-pregnant non-lactating females, 18 to 75 years of age (inclusive) at the time of screening.
* Body mass index (BMI) ≥18 and ≤35 (kg/m2), inclusive, and a minimum body weight of 45 kg.

Additional inclusion criteria might apply.

Exclusion Criteria:

* Symptoms consistent with COVID-19 such as fever, cough, and shortness of breath within 14 days before Day 1.
* Positive test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at screening or check-in (Day -1).
* Known previous COVID-19 infection.
* Use of any prescription or over-the-counter (OTC) medication, herbal products, or dietary supplements within the 7 days or 5 half-lives, whichever is longer, prior to the first study drug administration. Use of hormonal contraception is allowed prior to and during the study.

Additional exclusion criteria might apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Maximum measured concentration of total rilzabrutinib in plasma (Cmax) | Up to 48 hours after the last rilzabrutinib dose
Time from dosing to maximum measured concentration of total rilzabrutinib in plasma (tmax) | Up to 48 hours after the last rilzabrutinib dose
Area under the concentration-time curve of total rilzabrutinib in plasma from 0 to the last measurable concentration (AUC0-last) | Up to 48 hours after the last rilzabrutinib dose
Area under the concentration-time curve of total rilzabrutinib in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf) | Up to 48 hours after the last rilzabrutinib dose
Area under the plasma concentration-time curve of total rilzabrutinib from zero during the dosage interval (AUC0-tau) | Up to 48 hours after the last rilzabrutinib dose
Terminal Half-Life of total rilzabrutinib in Plasma (t1/2) | Up to 48 hours after the last rilzabrutinib dose
Apparent Total Clearance of rilzabrutinib in the plasma after oral administration (CL/F) | Up to 48 hours after the last rilzabrutinib dose
Apparent volume of distribution after oral administration (Vd/F) | Up to 48 hours after the last rilzabrutinib dose
Dose proportionality of rilzabrutinib | Up to 48 hours after the last rilzabrutinib dose
Accumulation ratio (Rac) | Up to 48 hours after the last rilzabrutinib dose

SECONDARY OUTCOMES:
Incidence of potentially clinically significant laboratory test, vital signs, and electrocardiogram (ECGs) abnormalities | Up to 14 days after rilzabrutinib dosing
Number of Adverse Events (AE) / Serious Adverse Events (SAE) | From date of signed ICF, up to 47 days
Bruton's Tyrosine Kinase (BTK) Occupancy characterization | Up to 48 hours after the last rilzabrutinib dose
Maximum measured concentration of rilzabrutinib metabolites in plasma (Cmax) | Up to 48 hours after the last rilzabrutinib dose
Time from dosing to maximum measured concentration of rilzabrutinib metabolites in plasma (tmax) | Up to 48 hours after the last rilzabrutinib dose
Area under the concentration-time curve of rilzabrutinib metabolites in plasma from 0 to the last measurable concentration (AUC0-last) | Up to 48 hours after the last rilzabrutinib dose
Area under the concentration-time curve of rilzabrutinib metabolites in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf) | Up to 48 hours after the last rilzabrutinib dose
Area under the plasma concentration-time curve of rilzabrutinib metabolites from zero during the dosage interval (AUC0-tau) | Up to 48 hours after the last rilzabrutinib dose
Terminal Half-Life of rilzabrutinib metabolites in Plasma (t1/2) | Up to 48 hours after the last rilzabrutinib dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number: 0001, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org